CLINICAL TRIAL: NCT01175525
Title: Treatment of Acute Stroke With Cromolyn(Single Dose)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Model: Parallel
Other Study IDs: 002
Record Dates: First submitted 2010-08-02; First posted 2010-08-05 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-08

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Cromolyn Sodium; Sugars

ARMS (2):
- sugar pill (Placebo Comparator): sugar pill dissolved in water to be given 4 times a day 30 minutes prior to meals
  Interventions: Drug: sugar pill
- Cromolyn (Active Comparator): Cromolyn dose of 200mg(dissolved in water) will be given 4 times a day(30 minutes before a meal)
  Interventions: Drug: CROMOLYN

INTERVENTIONS:
Drug: CROMOLYN — Cromolyn 200mg (dissolved in water) given 4 times a day
  Other Names: NASALCROM; GASTROCOM
  Arms: Cromolyn
Drug: sugar pill — sugar pill Dissolved in water taken 4 times daily 30 minutes prior to meals
  Arms: sugar pill

SUMMARY:
Mastocytes were proven to have a central rule in their development of the lipoid plaque of the vascular system. Mastocytes also has an important role in the stabilisation of the plaque in the building of the brain barrier. Different animal studies show that the inhibition of the mastocyte activity decreases significantly the risk of secondary bleeding post ischaemic stroke.It was also shown that post stroke inflammation process was also blocked by the inhibition of mastocytes.Other studies showed up to 100% decrease in the brain barrier disruption and post stroke oedema, after treatment with mastocyte inhibitors.

Cromolyn is a synthetic drug which has an anti-allergic effect by inhibition of the mastocytes. This drug is a well known,safe drug and is the main sub-substance that was used in the previously mentioned studies.

ELIGIBILITY:
Inclusion Criteria:

1. Infarction of the anterior Circulation system.
2. Both genders
3. Age > 20 years
4. NIHSS > 5 -

Exclusion Criteria:

1. Non- ischaemic stroke
2. Additional disease of the CNS
3. Known allergy to cromolyn
4. Diseae of mastocytosis
5. Renal or Hepatic failure (acute or chronic)
6. Inability to sign consent form (dementia or sensory aphasia)
7. Lacunar infarctions
8. INfarction present in cerebellum or brain stem -

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lampl, Neurologist, Principal Investigator — Wolfson Medical Center
Locations (1):
- Edith wolfson medical Center, Holon, Israel